CLINICAL TRIAL: NCT04533425
Title: Practical Approaches to Care in Emergency Syncope
Acronym: PACES
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marc Probst, Assistant Professor, Columbia University
Other Study IDs: AAAT5903; R01HL149680 (NIH); GCO 19-0127 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2020-08-27; First posted 2020-08-31 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Syncope; Presyncope
Keywords: Risk Score; Risk Stratification; External Validation
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for cardiac biomarker testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with syncope: Patients who present to the ED with syncope

SUMMARY:
Syncope, or transient loss of consciousness, is a common reason for visit to the Emergency Department and often leads to extensive testing and hospitalization. Using objective risk scores to determine which patients with syncope will actually benefit from these interventions, and which can be safely discharged home with minimal testing, is critical to providing sensible medical care. This study will evaluate the validity of two syncope risk-stratification tools and investigate their impact on healthcare utilization and patient safety, thus improving the quality of care for the 1-2 million patients who experience syncope every year in the United States

DETAILED DESCRIPTION:
The goal of this project is to improve risk-stratification for patients who present to the emergency department (ED) with syncope (transient loss of consciousness), in order to better delineate which patients require admission and which can be safely discharged home. Syncope and pre-syncope (the sensation of impending loss of consciousness) are common reasons to present to the ED, representing over 1.3 million visits per year in the United States.

Although syncope is most often benign, it can occasionally be caused by serious cardiopulmonary diseases such as cardiac arrhythmia, acute coronary syndrome, or pulmonary embolism. Despite thorough evaluation in the ED, the cause of syncope remains unknown in over 50% of cases, which leads to a large number of syncope patients being admitted for observation and/or further testing. These admissions to the hospital or observation unit are low-yield, costly, and expose patients to the possibility of iatrogenic harm.

In response to this, two groups of researchers have developed distinct syncope risk-stratification tools: the US Syncope Risk Score (FAINT) and the Canadian Syncope Risk Score. These scores use a combination of clinical, electrocardiographic, and laboratory variables to predict the risk of serious clinical outcomes at 30 days. While promising, these two risk scores require external validation prior to widespread clinical implementation. The study team will prospectively collect data on ~1,270 ED patients with syncope/pre-syncope and follow them for 30 days to validate the predictive accuracy of these two risk scores. The study team will then assess the impact of implementing these scores by measuring their potential effect on healthcare utilization and costs.

If validated and shown to safely reduce healthcare utilization, these syncope risk scores could play a major role in improving emergency syncope care by reducing low-yield admissions and identifying patients who are unsafe for discharge from the ED. This study, entitled PACES: Practical Approaches to Care in Emergency Syncope, will help increase the quality and value of emergency care, and advance the field of syncope research.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 40 years of age or older who present to the Emergency Department with syncope or presyncope.
* Subjects must read and speak English or Spanish.
* Subjects must have a working phone number and fixed address.

Exclusion Criteria:

* Patient who have a syncope mimic such as seizure, stroke, head trauma with loss of consciousness, altered mental status, hypoglycemia, intoxication, or require an intervention to restore consciousness.
* Patients who have a new serious diagnosis found in the Emergency Department, such as death, significant cardiac arrhythmia (see below), myocardial infarction, significant structural heart disease, stroke (both ischemic and hemorrhagic), pulmonary embolism, aortic dissection, hemorrhage or anemia requiring blood transfusion, subarachnoid hemorrhage, cardiopulmonary resuscitation, acute surgical illness, pregnancy, or major traumatic injury.
* Significant cardiac arrhythmia includes Ventricular Fibrillation, Ventricular tachycardia (>30 secs), Symptomatic ventricular tachycardia, (<30 secs), Sick sinus disease with alternating sinus bradycardia and tachycardia, Sinus pause > 3 seconds, Mobitz type II atrioventricular heart block, Complete heart block, Symptomatic supraventricular tachycardia (including Paroxysmal Supraventricular Tachycardia (PSVT), rapid atrial fibrillation/ flutter), Symptomatic bradycardia (pulse<40), Pacemaker or implantable cardioverter-defibrillator malfunction with cardiac pauses.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who presents to the Emergency Department (ED) after an episode of syncope or pre-syncope and who do not have a new serious diagnosis found during the index ED evaluation. There are no exclusions based on sex/gender, race, or ethnicity.
Sampling Method: Probability Sample
Enrollment: 1297 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
US Syncope Risk Score (The FAINT Score) | 30 days
  A combination of clinical, electrocardiographic, and laboratory variables to predict the risk of serious clinical outcomes at 30 days. Full scale range from 0-6, higher score indicates higher risk of a serious cardiac event or death.
Canadian Syncope Risk Score | 30 days
  A combination of clinical, electrocardiographic, and laboratory variables to predict the risk of serious clinical outcomes at 30 days. Full scale range from -3 to 11, higher score indicates higher risk of a serious clinical event or death.

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Probst, MD, MS, Principal Investigator — Columbia University
Locations (5):
- United States (5):
  - UC Davis, Sacramento, California
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Background] Probst MA, Kanzaria HK, Gbedemah M, Richardson LD, Sun BC. National trends in resource utilization associated with ED visits for syncope. Am J Emerg Med. 2015 Aug;33(8):998-1001. doi: 10.1016/j.ajem.2015.04.030. Epub 2015 Apr 24. PMID 25943042
- [Background] Probst MA, Gibson T, Weiss RE, Yagapen AN, Malveau SE, Adler DH, Bastani A, Baugh CW, Caterino JM, Clark CL, Diercks DB, Hollander JE, Nicks BA, Nishijima DK, Shah MN, Stiffler KA, Storrow AB, Wilber ST, Sun BC. Risk Stratification of Older Adults Who Present to the Emergency Department With Syncope: The FAINT Score. Ann Emerg Med. 2020 Feb;75(2):147-158. doi: 10.1016/j.annemergmed.2019.08.429. Epub 2019 Oct 23. PMID 31668571
- [Background] Thiruganasambandamoorthy V, Kwong K, Wells GA, Sivilotti MLA, Mukarram M, Rowe BH, Lang E, Perry JJ, Sheldon R, Stiell IG, Taljaard M. Development of the Canadian Syncope Risk Score to predict serious adverse events after emergency department assessment of syncope. CMAJ. 2016 Sep 6;188(12):E289-E298. doi: 10.1503/cmaj.151469. Epub 2016 Jul 4. PMID 27378464
- [Background] Wongtanasarasin W, Nishijima DK, Wood N, DeAngelis J, Storrow A, Schimmel J, Beltre N, Sacco D, Probst MA. Factors associated with incentive redemption among participants in a multicenter prospective syncope clinical study. Acad Emerg Med. 2024 Dec;31(12):1276-1279. doi: 10.1111/acem.14979. Epub 2024 Jun 28. No abstract available. PMID 38940329
- See also: Complete bibliography — https://www.ncbi.nlm.nih.gov/sites/myncbi/marc.probst.1/bibliography/47333221/public/?sort=date&direction=ascending